CLINICAL TRIAL: NCT00209599
Title: A Phase II, Randomized, Open-Label Study to Assess the Safety and Efficacy of AQUAVAN® Injection Versus Midazolam HCl for Sedation in Elderly Patients Undergoing Colonoscopy Procedures
Brief Title: A Study of AQUAVAN® Injection Versus Midazolam HCl for Sedation in Elderly Patients Undergoing Elective Colonoscopy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: PPD Development, LP (Industry); Covance (Industry); Quest Pharmaceutical Services (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3000-0415
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2008-11

CONDITIONS: Colonoscopy; Colon Polyps
Keywords: Colonoscopy; Seadation
MeSH Terms: conditions — Colonic Polyps | interventions — fospropofol

INTERVENTIONS:
Drug: fospropofol disodium

SUMMARY:
This study was designed to demonstrate that AQUAVAN® is effective in providing adequate sedation in elderly patients undergoing colonoscopy as well as to assess the safety profile of AQUAVAN versus that of midazolam. Prior to the procedure, patients received fentanyl citrate for pain management followed five minutes later by AQUAVAN® Injection for sedation. Throughout the procedure, study personnel assessed the patient's vital signs and depth of sedation. After the procedure, the patient, physician, and an evaluator were asked to complete satisfaction surveys.

DETAILED DESCRIPTION:
This is a randomized, open-label study designed to assess the safety and efficacy of AQUAVAN ® Injection versus midazolam HCl following pretreatment with an analgesic, fentanyl citrate injection, in producing sedation in elderly patients undergoing colonoscopy.

Following completion of preprocedure sedation assessments, patients will be randomly assigned to 1 of the 2 i.v. treatment groups at a 4:1 (AQUAVAN®. Injection: midazolam HCl) allocation ratio. To ensure that a distribution of ages is obtained, enrollment will be stratified into 2 equal-size groups by age (>65 to <72 years of age and >72 years of age). Randomization will be stratified by site within each age group. All patients will receive fentanyl citrate injection as an analgesic pretreatment. Supplemental doses of fentanyl citrate injection may be administered if the patient reports pain or if inadequate analgesia is present as demonstrated by increased heart rate and/or blood pressure in the presence of adequate sedation.

At no time should fentanyl citrate injection be administered to increase sedation levels.

AQUAVAN®. Injection and midazolam HCl will be administered to induce a state of adequate sedation, defined as a Modified Observer's Assessment of Alertness/Sedation (OAA/S) score of 4 or less. Supplemental doses will be administered to increase depth or duration of sedation. Supplemental doses will not be administered if the Modified OAA/S score is 2 or less or if there is no purposeful response to stimulation. The depth of sedation will be measured by the Modified OAA/S scale, a validated measure. Patient and Investigator assessments will be used to confirm the depth of sedation provided met the goals of sedation, reduction of anxiety and reduced awareness.

ELIGIBILITY:
Inclusion Criteria:

1. Patient provided a signed/dated Informed Consent and HIPAA authorization after receiving a full explanation of the extent and nature of the study.
2. Patient was over 65 years of age at the time of screening.
3. Patient met ASA Physical Status Classification of I to III.

Exclusion Criteria:

1. Patient had a history of allergic reaction or hypersensitivity to any anesthetic agent, narcotic, or benzodiazepine.
2. Patient did not meet nils per os (NPO) status per ASA Guideline or institution's guideline.
3. Patient had condition(s) that, in the opinion of the Investigator, could interfere with appropriate airway management.
4. Patient had a history of mental or visual impairment that would not permit successful measurement of cognitive evaluations.
5. Patient was unwilling to adhere to pre- and postprocedural instructions.
6. The use of fentanyl or midazolam was contraindicated for the patient.
7. Patient had participated in an investigational drug study within 1 month prior to study start.
8. Patient had prior exposure to AQUAVAN.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100
Dates: Start 2005-02; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint was Sedation Success defined as a patient having 3 consecutive Modified OAA/S scores ≤4 and completing the procedure without requiring alternative sedative medications and without requiring manual or mechanical ventilation.

SECONDARY OUTCOMES:
Measures of recovery and cognitive functions by the blinded evaluator
Time to Fully Recovered from the end of the procedure
Time to Fully Alert from the end of the procedure
Change from baseline DSST score over time during the Recovery period
Measures of sedation adequacy
Modified OAA/S scores over time during the Dosing Initiation, Procedural, and Recovery periods
Duration and percent of time when a patient's Modified OAA/S score is at each level between the first dose of study medication and Fully Alert, inclusive
Duration of sedation
Number of doses of study medication administered for the procedure
Time to sedation
Time that splenic flexure, hepatic flexure, and cecum are reached, and time to end of procedure
Number of repositionings
·Number of procedure interruptions due to inadequate sedation
Patient-reported outcome and Investigator's assessment
Patient's rating of experience after Fully Recovered (including patient's level of sedation, memory recall, pain/discomfort, and willingness to be treated again);
Patient's rating at 24-hour telephone survey (including time to normal food intake and time to resuming normal activities)
Investigator's rating at the end of the procedure (including patient's level of sedation, pain/discomfort, anxiety, response to instructions, overall satisfaction with the study drug, and willingness to be use sedatives again)
Blinded evaluator's rating after Fully Recovered
Safety Variables
The following were safety endpoints:
Nature, frequency, severity, relationship to treatment, and outcome of all treatment emergent AEs (TEAEs)
Airway management (manual repositioning, increased oxygen flow, verbal or tactile stimulation)
Airway intervention (suction, manual ventilation, endotracheal intubation or other mechanical airway management)
Sedation-related AEs (hypopnea, apnea, hypoxemia, bradycardia, hypotension,)
Alternative sedation/hypnotic medications

CONTACTS AND LOCATIONS:
Overall Officials: James Jones, MD,PharmD, Study Director — Eisai Inc.